CLINICAL TRIAL: NCT00006196
Title: The Relationship Between Vitamin D, Fingernail Thickness and Bone Density
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Diagnostic
Other Study IDs: NCRR-M01RR00036-0754; M01RR000036 (NIH)
Record Dates: First submitted 2000-09-07; First posted 2000-09-08 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Osteoporosis
Keywords: Vitamin D resistance
MeSH Terms: conditions — Osteoporosis | interventions — Vitamin D

INTERVENTIONS:
Drug: Vitamin D

SUMMARY:
Vitamin D deficiency is common in the elderly and contributes to the increased incidence of falls, hip fracture and depression in this population. An unknown number of elderly have vitamin D resistance resulting in a functional vitamin D deficiency state. Because there are no simple procedures or blood tests that identify vitamin D resistance, its prevalence and contribution to disability in the elderly is unknown. Our inability to screen for this condition precludes our ability to initiate and monitor treatment.

Previous studies indicate that fingernail thickness correlates with vitamin D status and may therefore provide a simple cost effective procedure to not only identify patients with vitamin D deficiency but also, those with vitamin D resistance. This procedure may also provide a way to monitor an individual's response to treatment.

This study is designed to demonstrate the association between fingernail thickness and vitamin D status.

ELIGIBILITY:
Inclusion Criteria:

* females 25-75 years of age with no known bone disorders

Exclusion Criteria:

* history of vertebral fractures or nonvertebral fractures without trauma
* prescription medications for prevention of osteoporosis (including vitamin D other than multivitamin and estrogen)
* history of malignancy other than basal cell or squamous cell cancer of the skin
* use of steroids or anticonvulsants in the 6 months prior to enrollment

Ages: 25 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- 4488 Forest Park, Suite 201, St Louis, Missouri, United States